CLINICAL TRIAL: NCT06592950
Title: Patient Preference Study in Type-2 Diabetes Mellitus: Discrete Choice Experiment (DCE) to Support Novo Nordisk's Long-Acting Insulin
Acronym: DCE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-7791; U1111-1293-3919 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Type-2 Diabetes Mellitus (T2DM)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Quantitative online survey: Across four markets (Canada, France, Spain and Japan)
  Interventions: Other: No treatment given
- Qualitative interviews: Conducted in Canada
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Online survey
  Groups: Quantitative online survey
Other: No treatment given — Interviews
  Groups: Qualitative interviews

SUMMARY:
The primary objective of this research is to assess T2DM patient preferences for a once weekly insulin treatment. The study involves a qualitative interview phase and quantitative survey phase with a Discrete Choice Experiment (DCE).

ELIGIBILITY:
Inclusion Criteria:

* Patient is an adult aged 18 years or over
* Patient was diagnosed with type-2 diabetes mellitus (T2DM) greater than or equal to 180 days prior to the day of screening
* Patient is currently prescribed a diabetes treatment (e.g., Metformin/Sus, DPP4i, SGLT2i, GLP-1 RA and/or basal insulin)
* Patient is willing and able to provide written informed consent to participate

For qualitative interviews:

* Patient is a fluent speaker of English and is able to read, write, and fully understand the English language
* Patient is a resident in Canada

For quantitative online survey:

* Patient is a fluent speaker of the local language (English/French/Spanish or Japanese) and is able to read, write and fully understand the local language
* Patient is a resident of either Canada, France, Spain or Japan

Exclusion Criteria:

* Patient is currently employing a basal-bolus insulin treatment regimen to manage their diabetes
* Patient is unwilling or unable to comply with the needs of the study or has a physical, behavioural or mental condition that, in the opinion of the recruiter may affect the patient's ability to take part in the study, understand the nature, scope and possible consequences of the study, or the responses they might provide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type-2 diabetes mellitus (T2DM) patients
Sampling Method: Non-Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
T2DM patient preferences for a once weekly insulin treatment | Day of interview/survey completion (Day 1)
  Pre-defined open-ended questions and Discrete Choice Experiment online survey

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk, Søborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com